CLINICAL TRIAL: NCT00215111
Title: Role of Carbohydrate Modification in Weight Management Among Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Shelley Kirk, Ph.D., R.D., L.D., Associate Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02819-8
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Childhood Obesity
Keywords: childhood obesity; weight management; dietary interventions; cardiovascular disease risk factors
MeSH Terms: conditions — Pediatric Obesity

ARMS (1):
- Low carbohydrate, reduced glycemic load, control diet (Experimental)
  Interventions: Behavioral: Low carbohydrate, reduced glycemic load, and a control diet

INTERVENTIONS:
Behavioral: Low carbohydrate, reduced glycemic load, and a control diet

SUMMARY:
The purpose of this study is to test the hypothesis that a low-carbohydrate diet and a low-glycemic load diet will improve body mass index and result in more body fat loss than a control diet among overweight children ages 7 to 12. In addition this study is also designed to test the safety of diets with modified carbohydrate content as compared to a conventional weight management diet among younger overweight children.

DETAILED DESCRIPTION:
The treatment of pediatric obesity supported by the medical community is a moderate restriction in calories by modifying intake of fat and simple sugars, along with an increase in energy expenditure through more physical activity. However, this approach is associated with only limited success. As a result, overweight children and adolescents are seeking alternative approaches to weight management, such as diets that modify the type and amount of carbohydrates. However, at this time there is limited data on the safety and efficacy of these diets, particularly with younger children. This study is a controlled clinical trial that compares the safety and efficacy of a low carbohydrate and reduced glycemic load diets to a more standard dietary intervention for the management of pediatric obesity (i.e. portion-controlled, moderate fat, high carbohydrate diet). This study will involve 150 overweight children (ages 7 to 12) who will be randomly assigned to one of the three diet groups for 12 months. The effects of each diet will be determined by measuring changes in anthropometric measures (body weight, height, body mass index, waist circumference, body composition), other cardiovascular risk factors (blood pressure, fasting lipid profile, fasting glucose and insulin, and inflammatory markers of cardiovascular disease), and measures of psychological well-being and mental status. The results of this study will provide needed information to the public in their quest for safe, effective, and health-promoting weight management strategies for obese children. Such information is vital if we are to address the obesity epidemic in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-12 years
* Body mass index >95th percentile and BMI z-score no greater than 2.65
* Normal fasting blood glucose of less than 100 mg/dL
* Age-appropriate cognitive and behavioral skills
* Absence of developmental or physical disabilities
* Capability to function independently in group exercise sessions
* Commitment of parent/guardian to attend scheduled meetings for 12-month period

Exclusion Criteria:

* Active cardiac, pulmonary, renal, liver, or gastrointestinal disease (pancreatitis, cholelithiasis, inflammatory bowel disease), diabetes, untreated thyroid disease, hypertension, hyperlipidemia
* Chronic infections
* Uncompensated or labile mental illness
* Chronic or intermittent use of corticosteroids
* Specific medications that may alter lipid, glucose, bone metabolism or appetite

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2005-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The outcomes listed below will be obtained at baseline,3-month, | 3 month
6-month and 12-month assessments unless otherwise noted,body weight, | 6-month and 12-month
height,body mass index,waist circumference,percent body fat, | baseline, 3-month, 6-month and 12-month
adipose mass,lean body mass,bone mineral density,fasting lipid profile, | baseline, 3-month, 6-month and 12-month
fasting insulin,fasting glucose,2-hour glucose (baseline and 3-month assessment), | baseline, 3-month, 6-month and 12-month

SECONDARY OUTCOMES:
physical activity (3-day physical activity records and pedometer readings) | 3-month, 6-month and 12-month
compliance with behavioral intervention (frequency rewards were earned) | weekly
attendance at group and individual sessions during initial 3-month intervention | 3-month, 6-month and 12-month
Sexual Maturity Rating | baseline
Hunger/Satiety assessment (Three-Factor Eating Questionnaire) | baseline, 3-month, 6-month and 12-month
Parent/guardian perception of success for each diet assignment prior to their child being randomized to a diet group | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Shelley Kirk, Ph.D., R.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States